CLINICAL TRIAL: NCT06059989
Title: A Multicenter Randomized, Open-label Study to Compare the Efficacy of Subcutaneous Infliximab Monotherapy with Subcutaneous Infliximab and Concomitant Immunosuppression in the Treatment of Moderate to Severe Crohn's Disease
Brief Title: InDuctIon TREatment with SubCuTaneous Infliximab for Crohn's Disease
Acronym: DIRECTCD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Principal Investigator, Krisztina Gecse, Medical Docter IBD specialist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL76663.018.21
Record Dates: First submitted 2023-03-13; First posted 2023-09-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Disease; Disease Crohn; Bowel Disease
Keywords: Crohn's disease; Biological; Subcutaneous
MeSH Terms: conditions — Crohn Disease; Intestinal Diseases | interventions — CT-P13; Immunosuppressive Agents; Mercaptopurine; Methotrexate; Folic Acid

STUDY DESIGN:
Intervention Model Description: Prospective Multicenter Randomized Controlled, Open-label Non-inferiority Study to Investigate the Efficacy of Subcutaneous Infliximab with and without Immunomodulators during Induction treatment in Moderate to Severe Crohn's Disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monotherapy (Experimental): Group 1: Monotherapy group
  Patients randomized to IFX monotherapy start with subcutaneous IFX 240mg at week 0 and 2 and then from week 4, 120mg s.c.EOW.
  Interventions: Drug: Infliximab subcutaneous
- Combination therapy (Experimental): Group 2: Combination therapy group
  Patients randomized to IFX combination therapy start with subcutaneous IFX 240mg at week 0 and 2 and then from week 4, 120mg s.c. EOW.
  Patients randomized to IFX combination therapy also receive Immunosuppressives EOW.
  Interventions: Drug: Infliximab subcutaneous; Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Infliximab subcutaneous — Mono and combination therapy group
  Other Names: Remsima 120mg solution s.c.
Drug: Immunosuppressive Agents — Combination group only
  Other Names: 6-mercaptopurine 1-1.5 mg/kg oral; or, if already on oral azathioprine or thioguanine continuous dosing 2-2.5mg/kg, or 20mg once daily respectively; In case of adverse events or investigator's individual consideration, instead of thiopurine, methotrexate 15 mg/week s.c. (or oral) in combination with oral folic acid 5 mg/week
  Arms: Combination therapy

SUMMARY:
Study Design:

A Prospective Multicenter Randomized Controlled, Open-label Non-inferiority Study to Investigate the Efficacy of Subcutaneous (SC) Infliximab (IFX) with and without Immunomodulators during Induction treatment in Moderate to Severe Crohn's Disease.

Primary endpoint:

The proportion of patients in corticosteroid-free clinical remission (as defined by a Crohn's disease activity index (CDAI)<150) and endoscopic response (as defined by a simple endoscopic score for Crohn's disease (SES-CD) drop of at least 50%) at week 26.

Accrual and feasibility:

This study will enroll 158 subjects at approximately 20 sites in the Netherlands (peripheral and academic hospitals). The estimated enrollment is 0.5 patient/centre/month leading to an inclusion duration of 16 months once all centres are open. The first enrolment is anticipated in Q1 2021.

Treatment, dosage and administration:

Eligible patients will be randomized to receive SC IFX monotherapy (240mg at week 0 and week 2 and then 120mg every other week (EOW) OR SC IFX (240mg at week 0 and week 2 and then 120mg EOW) in combination with immunosuppression.

DETAILED DESCRIPTION:
Permitted concomitant medications:

Oral prednisone (≤40 mg per day) or budesonide (≤9 mg per day) are permitted if on stable dose 2 weeks prior to screening. After 2 weeks into treatment, systemic corticosteroids will be tapered at a rate of at least 5 mg per week and budesonide will be tapered at a rate of 3 mg every 2 weeks. If tapering fails, re-introduction of lowest effective dose of corticosteroid is allowed a single time at the discretion of the treating physician, after which tapering is required beginning 2 weeks later.

Stable doses of mesalazine (at a maximum dose of 4g/day) are permitted throughout the study.

Stable doses of antibiotics are permitted until week 12. Adverse events to antibiotics can prompt treatment discontinuation, in that case a switch is allowed during week 12.

Patients randomized to IFX combination therapy will also receive 6-mercaptopurine 1-1.5 mg/kg. If participants are already using azathioprine or thioguanine, they will receive continued dosing 2-2.5mg/kg or 20mg once daily, respectively (unless shunter status or previous adverse events suggest differently). In case of previous adverse event leading to thiopurine discontinuation methotrexate 15 mg/week sc. in combination with oral folic acid 5mg/week will be prescribed.

Immunosuppressive treatment will be stopped at screening (approximately 2 weeks before randomization) for all patients and will be restarted for patients in the combination treatment group. Patients randomized to IFX monotherapy will not receive concomitant immunosuppression.

Primary Objectives:

The aim of this study is to investigate the efficacy of subcutaneous IFX in the treatment of moderate to severe Crohn's disease with and without concomitant immunosuppression, as measured by the proportion of patients in corticosteroid-free clinical remission (as defined by a CDAI<150) and endoscopic response (as defined by a SES-CD drop of at least 50%) at week 26. The Investigator hypothesizes that subcutaneous IFX monotherapy is non-inferior to subcutaneous IFX with concomitant immunosuppression in inducing this combined primary endpoint of corticosteroid free remission (CSF), clinical remission and endoscopic response by week 26.

Secondary Objectives: (not hierarchical)

* The proportion of patients in endoscopic remission at week 26 (defined as the absence of ulcerations larger then 5mm)
* Proportion of patients with endoscopic remission at week 26 (as measured by SES-CD≤2)
* Proportion of patients with endoscopic response at week 26 (as measured by at least 50% reduction in the SES-CD as compared to baseline)
* Proportion of patients in corticosteroid-free clinical remission at week 26 (defined as a CDAI<150)
* The proportion of patients in corticosteroid-free remission (CSF) deep remission at week 26, as defined by corticosteroid-free clinical (CDAI<150) AND endoscopic remission (defined as the absence of ulcerations larger then 5mm)
* Proportion of patients in clinical remission at week 2, 4, 8, 14 and 26 (defined as a CDAI<150)
* Proportion of patients achieving clinical response at week 2, 4, 8, 14 and 26 (defined as a CDAI-70)
* Proportion of patients achieving clinical response at week 26 (defined as a CDAI-100)
* Proportion of patients in symptomatic remission at week 2, 4, 8, 14 and 26 (defined as a patient reported outcome (PRO-2) (stool frequency and abdominal pain) <8)
* Proportion of patients achieving symptomatic response at week 2, 4, 8, 14 and 26 (defined as a PRO-2 -8)
* Time to symptomatic remission (defined as a PRO-2 (stool frequency and abdominal pain) <8)
* Proportion of patients in biochemical remission at week 8, 14 and 26 : C-reactive protein (CRP ≤ 5.0 mg/L and fecal calprotectin < 250 mg/g)
* Time to biochemical remission (CRP ≤ 5.0 mg/L and fecal calprotectin < 250 mg/g)
* Proportion of patients achieving minimally clinically important difference in quality of life at week 2, 4, 8, 14 and week 26 compared to baseline as assessed by the inflammatory bowel disease questionnaire (IBDQ) and EuroQol - 5 dimension - 5 level (EQ-5D-5L) questionnaire
* Proportion of patients developing anti-drug antibodies (ADA) against IFX at week 2, 4, 8, 14 and 26 as measured by a drug-tolerant assay
* IFX trough levels at week 2, 4, 8, 14 and 26
* Human Leukocyte antigen (HLA) haplotyping and correlation with anti-drug antibodies (ADA) development
* Thiopurine metabolites at baseline, week 14 and week 26 (for patients randomized for the combination therapy group, only at baseline for those in the monotherapy group and with previous IS use)
* Proportion of patients having IFX trough levels of >5ug/ml at week 26
* Proportion of patients achieving histological healing at week 26
* Proportion of patients (of those with active perianal disease at baseline) in clinical remission and response of their perianal disease, as defined by the fistula drainage assessment at week 26
* Proportion of patients with extraintestinal manifestations at week 26 as compared to baseline
* Adverse events.

Subject Population:

158 patients with moderate to severe Crohn's disease between the age of 18-80 years who are starting with IFX treatment.

Treatment Arms:

Group 1: Subcutaneous IFX monotherapy 240mg at week 0 and week 2 and then 120mg EOW.

Group 2: Subcutaneous IFX 240mg at week 0 and week 2 and then 120mg EOW in combination with immunosuppressive.

Randomly assigned to either of these groups in a 1:1 ratio. Randomization will be stratified according to immunosuppressive use at screening.

Duration of Treatment: 26 weeks. Period of evaluation: 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older diagnosed with Crohn's disease
2. Patients with moderate to severely active Crohn's disease with a Crohn's Disease Activity Index (CDAI) of 250 to 450 and presence of endoscopic ulceration in the terminal ileum, colon or both. Minimal SES-CD is ≥ 6 or ≥ 4 for isolated ileal disease.
3. Patients who had no response or loss of response to or have had intolerable side effects to one or more to the following: glucocorticoids, thiopurines (azathioprine/6-mercaptopurine/6-thioguanin), methotrexate , adalimumab, vedolizumab or ustekinumab OR patients in need of immediate top-down treatment with IFX at the discretion of the treating physician.
4. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
5. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedure.
6. Male or non-pregnant, non-lactating females. No wish to become pregnant in the coming 26 weeks.

Exclusion Criteria:

1. Patients at imminent need of surgery as judged by the treating clinician
2. Patients with the short bowel syndrome, an ostomy or a symptomatic non-inflammatory stricture
3. Patients previously exposed to IFX (intravenous or subcutaneous)
4. Previously unacceptable side effects or intolerance to all immunosuppressants (both thiopurines and methotrexate)
5. Treatment with adalimumab or vedolizumab or ustekinumab within 30 days
6. Patients who have had a primary non-response to adalimumab or had intolerable class-related side effects (as evaluated at the discretion of the treating physician)
7. Enteric pathogens (such as Salmonella, Shigella, Yersinia, Campylobacter and C. difficile) detected by stool analysis within 2 weeks prior to enrollment or at screening
8. Ongoing participation in another interventional trial
9. Patients with Ulcerative Colitis or Inflammatory bowel disease unclassified (IBD-U)
10. Patients with ongoing abdominal or undrained perianal abscess
11. Patients with a history of colon cancer or colonic dysplasia, unless sporadic adenoma, which has been removed
12. Active or latent tuberculosis (screening according to national guidelines). Except when the latter has been treated appropriately according to national guidelines.
13. Cardiac failure in the New York heart Association (NYHA) stage III-IV
14. History of demyelinating disease
15. Recent live vaccination (≤ 4 weeks)
16. Patients with ongoing acute/chronic infection (including but not limited to HIV, hepatitis B and C) with the exception of chronic herpes labialis or cervical human papillomavirus (HPV)
17. History of cancer in the last 5 years with the exception of non-melanoma skin cancer
18. Male patients with Epstein-Barr virus (EBV) negative serology
19. A history of alcohol or illicit drug use that in the opinion of the principal investigator (PI) would interfere with study procedures
20. Patients with psychiatric problems that in the opinion of the PI would interfere with study procedures
21. Patients unable to attend all study visits
22. Patients with a history of non-compliance with clinical study protocols
23. Contraindication for endoscopy
24. Patients who received any investigational drug in the past 30 days or 5 half-lives, whichever is longer
25. Pregnancy or lactation or wish to become pregnant in the coming 26 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Crohn's disease activity index <150 (-10 to 480) AND endoscopic response , where the higher score means worse outcome . | at week 0 and 26
  The proportion of patients in corticosteroid-free clinical remission.

SECONDARY OUTCOMES:
Endoscopic remission | week 0 and 26
  The proportion of patients with absence ulcerations larger then 5mm
Simple Endoscopic score for Crohn's disease ≤2 ( 0-60) where a higher score means worse outcome | week 0 and 26
  Proportion of patients with endoscopic remission
Crohn's disease activity index <150 (-10 to 480) where a higher score is a worse outcome | week 0, 2, 4, 8, 14 and 26
  Number of patients in clinical remission
Crohn's disease activity index improved with 70 points (-10 to 480) where a higher score is a worse outcome. | week 0, 2, 4, 8, 14 and 26
  Proportion of patients achieving clinical response
Crohn's disease activity index improved by100 points( -10 to 480) where a higher score is a worse outcome | at week 26
  Proportion of patients achieving clinical response
Patient reported outcome PRO-2 (stool frequency and abdominal pain) <8 (0 to na) where the higher score is the worse outcome | week 0, 2, 4, 8, 14 and 26
  Proportion of patients in symptomatic remission
CRP ≤ 5.0 mg/L | at week 0 and 4, 8, 14 and week 26
  Proportion of patients in biochemical remission
Inflammatory bowel disease questionnaire | at week 0, 2, 4, 8, 14 and week 26
  Proportion of patients achieving minimally clinically important difference in quality of life
Drug-tolerant assay | week 2, 4, 8, 14 and 26
  Proportion of patients developing anti-drug antibodies (ADA) against IFX
Thiopurine metabolites test | At baseline, week 14 and week 26 (for patients randomized for the combination therapy group. Only at baseline for those in the monotherapy group and with previous IS use)
  Level of Metabolites 6mmp, 6-tgn
IFX concentrate levels | week 2, 4, 8, 14 and 26
  IFX trough levels of > 5ug/ml at week 26
Histological analysis | week 0 and week 26
  Proportion of patients achieving histological healing
Fistula drainage assessment | week 0 and week 26
  Proportion of patients (of those with active perianal disease at baseline) in clinical remission and response of their perianal
Number of adverse event reports | week 0 to week 26
  Number of adverse event recorded in mono and combination therapy group
EuroQol-5Dimension-5Level questionnaire | at week 0, 2, 4, 8, 14 and week 26
  Proportion of patients achieving minimally clinically important difference in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dr. G D'Haens, Phd MD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No